CLINICAL TRIAL: NCT02451930
Title: An Open-Label, Multicenter, Phase 1b Study With an Expansion Cohort to Evaluate Safety and Efficacy of the Combination of Necitumumab With Pembrolizumab in Patients With Stage IV Non-Small Cell Lung Cancer
Brief Title: A Study of the Combination of Necitumumab (LY3012211) and Pembrolizumab (MK3475) in Participants With NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15568; I4X-MC-JFCQ (Other: Eli Lilly and Company); 2015-001291-22 (EudraCT Number); KEYNOTE -099 (Other: Merck)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2019-10-01

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — necitumumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Necitumumab + Pembrolizumab (Experimental): Part A Cohort 1: 600 mg Necitumumab + 200 mg Pembrolizumab:
  Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 600 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC (all histologies).
  Part A Cohort 2, Part B and Part C: 800mg Necitumumab + 200mg Pembrolizumab:
  Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part A cohort 2 participants with any histology, Part B and C participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japan participants. Part C were Japan participants.
  Interventions: Drug: Necitumumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: LY3012211
Drug: Pembrolizumab — Administered IV
  Other Names: MK3475

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the combination of necitumumab with pembrolizumab in participants with stage IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* The participant has Stage IV NSCLC.

  * Part A: NSCLC Stage IV (any type)
  * Part B: NSCLC Stage IV (squamous and nonsquamous)
  * Part C: NSCLC Stage IV in Japanese participants (squamous and nonsquamous)
* The participant must have progressed after 1 platinum-based chemotherapy regimen for Stage IV NSCLC. Prior therapy with VEGF/VEGFR targeting agents is permitted. Prior neoadjuvant/adjuvant therapy is permitted. Prior treatment with EGFR-TKI and ALK inhibitors is mandatory in participants with NSCLC whose tumor has EGFR-activating mutations or ALK translocations, respectively.
* Measurable disease at the time of study entry as defined by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1).
* The participant has evaluable tumor tissue available for biomarker analyses.
* The participant has adequate organ function.
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0-1.

Exclusion Criteria:

* The participant is currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 monoclonal antibody.
* Have a serious concomitant systemic disorder or significant cardiac disease.
* The participant has undergone major surgery or received anti-cancer monoclonal antibody therapy in the 30-days prior to study enrollment.
* The participant has undergone chest irradiation within 2 weeks prior to receiving study treatment.
* The participant has brain metastases that are symptomatic.
* The participant has a history of arterial thromboembolism event (ATE) or venous thromboembolism event (VTE) within 3 months prior to study enrollment. Participants with history of VTE beyond 3 months prior to study enrollment can be enrolled if they are appropriately treated with low molecular weight heparin.
* The participant has a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab or pembrolizumab, or any other contraindication to one of the administered treatments.
* The participant has a concurrent active malignancy. Previous history of malignancy is permitted, provided that the participant has been free of disease for ≥3 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, preinvasive carcinoma of the cervix, or any cancers that in the judgment of the investigator and sponsor may not affect the interpretation of results (for example, prostate, bladder).
* History of interstitial lung disease, pneumonitis, autoimmune disease or syndrome that requires steroids or immunosuppressive agents.
* The participant has active infection requiring systemic therapy, including active tuberculosis or known history of infection with the human immunodeficiency virus (HIV 1/2 antibodies), or hepatitis B (e.g., HBsAg reactive) and/or C virus (e.g., HCV RNA [qualitative] is detected).
* The participant has an active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* The participant has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (3):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Tennessee Oncology PLLC, Nashville, Tennessee
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sunto-Gun
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: A Study of the Combination of Necitumumab (LY3012211) and Pembrolizumab (MK3475) in Participants With NSCLC — http://www.lillytrialguide.com/en-US/studies/non-small-cell%20lung%20cancer/JFCQ#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, participants in Part A Cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Groups:
- Part A Cohort 1: 600 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab (pembro) absolute dose by intravenous (IV) infusion on Day1 of 21 days cycles followed by 600 mg necitumumab (Neci) absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC (all histologies).
- Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part A cohort 2 participants with any histology, Part B and C participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japan participants.
Period: Overall Study
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro
Started | 3 | 68
Received at Least One Dose of Study Drug | 3 | 68
Part A Cohort 2 Participants | 0 | 6
Part B Participants | 0 | 55
Part C Participants | 0 | 7
Completed | 1 | 38
Not Completed | 2 | 30
Not completed — Death | 0 | 15
Not completed — Lost to Follow-up | 0 | 3
Not completed — Sponsor Decision | 2 | 10
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Groups:
- Part A Cohort 2 and Part B: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC of squamous and nonsquamous histology.
- Part C: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japan participants.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2 and Part B: 800 mg Neci + 200 mg Pembro | Part C: 800 mg Neci + 200 mg Pembro | Total
Number analyzed (Participants) | 3 | 61 | 7 | 71
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part A and B | 67.0 (7.21) | 63.13 (9.82) | NA (NA) — This row represents Part A and Part B data only. | 63.31 (9.73)
  Part C | NA (NA) — This row represents Part C data only. | NA (NA) — This row represents Part C data only. | 64.14 (8.55) | 64.14 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 17 | 2 | 20
  Male | 2 | 44 | 5 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 21 | 0 | 22
  Unknown or Not Reported | 2 | 39 | 7 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 7 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 3 | 47 | 0 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 13 | 0 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 7 | 0 | 7
  Japan | 0 | 0 | 7 | 7
  France | 2 | 40 | 0 | 42
  Spain | 1 | 14 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Part A and Part C
Description: A dose limiting toxicity (DLT) was defined as an adverse event (AE) during the first 21 days that was possibly related to the study drug and fulfilled any of the following criteria using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0: Grade 3 or 4 nonhematologic toxicity, Grade 4 nausea, vomiting, or diarrhea that persists more than 3 days despite maximal supportive intervention, Grade 3 thrombocytopenia with bleeding requiring transfusion, Grade 4 thrombocytopenia with or without bleeding, Grade 4 neutropenia that persists more than 5 days, Grade 3 or 4 neutropenia with fever, Grade ≥3 skin toxicity despite best supportive care with some exceptions, if a total at least 75% of the planned dose for both agents cannot be administered in the first cycle due to toxicity, prolonged delay (>2 weeks) in initiating cycle 2 due to treatment-related toxicity and Grade 5 toxicity.
Time Frame: Baseline through Cycle 1 (21 day cycles)
Population: All participants who received at least one dose of study drug in Part A and Part C.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort 2: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC (all histologies).
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2: 800 mg Neci + 200 mg Pembro | Part C: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 3 | 6 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) (Objective Response Rates [ORR]) in Part A and Part B
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Up To 16 Months)
Population: All participants who received at least one dose of study drug in Part A and Part B. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part B participants with Stage IV NSCLC of squamous and nonsquamous histology and Part A cohort 2 participants with all histologies.
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 3 | 61
Percentage of Participants | 66.7 [9.4 to 99.2] | 21.3 [11.9 to 33.7]
Statistical Analysis 1: Comparison: Part A Cohort 1: 600 mg Neci + 200 mg Pembro vs Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro; Test type: Other; p = 0.4491, Fisher Exact

3. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR) (Objective Response Rates [ORR]) in Part A Cohort 2, Part B and Part C
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Up To 40 Months)
Population: All participants who received at least one dose of study drug in Part A Cohort 2, Part B and Part C. Part C were Japan participants. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A Cohort 2, Part B and Part C: 800 mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part A cohort 2 participants with any histology, Part B and C participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japan participants.
Arm/Group | Part A Cohort 2, Part B and Part C: 800 mg Neci + 200mg Pembro
Number analyzed (Participants) | 68
percentage of participants | 25.0 [15.3 to 37]

4. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab in Part A, Part B and Part C
Description: Pharmacokinetics (PK): Minimum Concentration (Cmin) of Necitumumab.
Time Frame: Predose sample (within 1 hour before infusion) and postdose sample (within 10 min after infusion) on Day 1 at Cycles 1, 2, 4, 6, 8; 30 days post treatment discontinuation
Population: All participants who received at least one dose of study drug and had evaluable PK data in Part A, Part B and Part C.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- Part B: 800mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC of squamous and nonsquamous histology.
- Part C: 800mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japanese participants.
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2: 800 mg Neci + 200 mg Pembro | Part B: 800mg Neci + 200mg Pembro | Part C: 800mg Neci + 200mg Pembro
Number analyzed (Participants) | 3 | 6 | 44 | 7
micrograms per milliliter (μg/mL)
  Pre-Dose Cycle 2: number analyzed (Participants) | 3 | 6 | 43 | 5
  Pre-Dose Cycle 2 | 50.4 (54.7) | 70 (49.7) | 58.2 (56) | 90.4 (18.4)
  Pre-Dose Cycle 4: number analyzed (Participants) | 3 | 3 | 35 | 4
  Pre-Dose Cycle 4 | 79.2 (32.5) | 148 (32.1) | 101 (48) | 136 (9.51)
  Pre-Dose Cycle 6: number analyzed (Participants) | 3 | 3 | 28 | 3
  Pre-Dose Cycle 6 | 89.5 (24.7) | 195 (12.2) | 114 (58.3) | 114 (66.5)
  Pre-Dose Cycle 8: number analyzed (Participants) | 3 | 2 | 21 | 3
  Pre-Dose Cycle 8 | 98.5 (3.73) | 155 (33) | 91 (62.7) | 209 (18.7)
  End-of-Infusion Cycle 1 | 152 (32.1) | 269 (15.6) | 226 (24.6) | 281 (26)
  End-of-Infusion Cycle 2: number analyzed (Participants) | 3 | 6 | 36 | 5
  End-of-Infusion Cycle 2 | 194 (29) | 352 (25.3) | 273 (36.8) | 391 (25.4)
  End-of-Infusion Cycle 4: number analyzed (Participants) | 3 | 4 | 31 | 4
  End-of-Infusion Cycle 4 | 246 (28.7) | 353 (45.3) | 315 (45.4) | 428 (5.18)
  End-of-Infusion Cycle 6: number analyzed (Participants) | 3 | 3 | 24 | 3
  End-of-Infusion Cycle 6 | 234 (26.3) | 396 (8.53) | 312 (42.1) | 406 (12.9)
  End-of-Infusion Cycle 8: number analyzed (Participants) | 3 | 2 | 17 | 2
  End-of-Infusion Cycle 8 | 291 (20.8) | 526 (8.49) | 295 (46.4) | 507 (7.95)

5. Secondary Outcome: Number of Participants With Anti-Necitumumab Antibodies in Part A, Part B and Part C
Description: Result is considered as treatment emergent anti-necitumumab antibody positive if postbaseline titer = 4*baseline titer for baseline titer > 0 or if postbaseline titer >= 20 for samples with antibody not detected.
Time Frame: Predose Cycle 1 Day 1 through Predose Cycle 8 Day 1 (21 Day Cycles)
Population: All participants who received at least one dose of study drug who had evaluable data in Part A, Part B and Part C.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort 1: 600mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab (pembro) absolute dose by intravenous (IV) infusion on Day1 of 21 days cycles followed by 600 mg necitumumab (Neci) absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC (all histologies).
- Part A Cohort 2 and Part B: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part B participants with Stage IV NSCLC of squamous and nonsquamous histology and Part A cohort 2 participants with all histologies.
- Part C: 800 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 every 21 days followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21-day cycles in participants with Stage IV NSCLC of squamous and nonsquamous histology.
  Part C were Japan participants.
Arm/Group | Part A Cohort 1: 600mg Neci + 200mg Pembro | Part A Cohort 2 and Part B: 800 mg Neci + 200 mg Pembro | Part C: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 3 | 61 | 7
Participants | 0 | 2 | 0

6. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), and Stable Disease (SD) (Disease Control Rate [DCR]) in Part A Cohort 2 and Part B
Description: Disease control rate (DCR) is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Up To 16 Months)
Population: All participants who received at least one dose of study drug in Part A Cohort 2 and Part B. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 61
percentage of participants | 62.3

7. Secondary Outcome: Duration of Response (DoR) in Part A Cohort 2 and Part B
Description: DOR was defined only for responders (participants with confirmed CR or PR). It was measured from the date of first evidence of a confirmed CR or PR to the date of objective progression or the date of death due to any cause, whichever was earlier.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up To 16 Months)
Population: All participants who received at least one dose of study drug who had evaluable data in Part A Cohort 2 and Part B. 11 participants were censored. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 4
months | 10.94 [4.17 to NA] — Upper confidence interval was not evaluable due to high censoring.

8. Secondary Outcome: Progression Free Survival (PFS) in Part A Cohort 2 and Part B
Description: PFS was defined as the time from the date of first dose of study drug until first observation of objective (radiographically documented) PD as defined by RECIST v1.1 or death from any cause, whichever comes first. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Death Due to Any Cause (Up To 16 Months)
Population: All participants who received at least one dose of study drug and who had evaluable data in Part A Cohort 2 and Part B. 21 participants were censored. Per protocol, participants in Part A cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Cohort 2 and Part B: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 40
Months | 3.98 [2.23 to 6.87]

9. Secondary Outcome: Overall Survival (OS) in Part A Cohort 2, Part B
Description: OS duration was measured from the date of first dose of study drug (necitumumab and/or pembrolizumab) to the date of death from any cause.
Time Frame: Baseline to Death from Any Cause (Up To 16 Months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A Cohort 2, Part B: 800 mg Neci + 200 mg Pembro
Number analyzed (Participants) | 61
months | NA [NA to NA] — OS was not reached because data were not mature at data cutoff.

ADVERSE EVENTS:
Time Frame: Baseline Up to 49 Months
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At risk adjusted accordingly. Per protocol, participants in Part A Cohort 2 who received the recommended necitumumab dose for Part B were also analyzed together with Part B.
Groups:
- Part A Cohort 1: 600 mg Neci + 200 mg Pembro: Participants received 200 mg pembrolizumab (pembro) absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 600 mg necitumumab (Neci) absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in participants with Stage IV NSCLC (all histologies).
- Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro: Participants received 200 mg pembrolizumab absolute dose by intravenous (IV) infusion on Day 1 of 21 days cycles followed by 800 mg necitumumab absolute dose by IV infusion on Days 1 and 8 of 21 days cycles in Part B and C participants with Stage IV NSCLC of squamous and nonsquamous histology and Part A cohort 2 participants with any histology.
  Part C were Japan participants.
Arm/Group | Part A Cohort 1: 600 mg Neci + 200 mg Pembro | Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro
All-Cause Mortality (participants affected / at risk) | 0/3 | 23/68
Serious Adverse Events (participants affected / at risk) | 1/3 | 30/68
Other Adverse Events (participants affected / at risk) | 3/3 | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: 600 mg Neci + 200 mg Pembro (N=3) | Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro (N=68)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (4)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Fixed eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A Cohort 1: 600 mg Neci + 200 mg Pembro (N=3) | Part A Cohort 2, Part B and Part C: 800mg Neci + 200mg Pembro (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 7 (11)
Hypothyroidism (Endocrine disorders) | 1 (1) | 5 (7)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 11 (16)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 16 (23)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (13)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (5) | 16 (26)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (17)
Asthenia (General disorders) | 1 (1) | 22 (46)
Chills (General disorders) | 0 (0) | 5 (5)
Fatigue (General disorders) | 1 (3) | 21 (29)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (3)
Oedema peripheral (General disorders) | 1 (1) | 5 (6)
Pyrexia (General disorders) | 1 (1) | 9 (21)
Xerosis (General disorders) | 0 (0) | 8 (28)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 8 (10)
Folliculitis (Infections and infestations) | 0 (0) | 5 (10)
Paronychia (Infections and infestations) | 2 (3) | 10 (18)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5)
Skin infection (Infections and infestations) | 1 (1) | 7 (11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 11 (17)
Amylase increased (Investigations) | 0 (0) | 4 (19)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 10 (21)
Blood alkaline phosphatase increased (Investigations) | 1 (4) | 7 (9)
Blood creatine phosphokinase increased (Investigations) | 1 (4) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 6 (7)
International normalised ratio increased (Investigations) | 1 (3) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 4 (22)
Weight decreased (Investigations) | 0 (0) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 20 (26)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (12) | 24 (62)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 9 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7)
Dizziness (Nervous system disorders) | 0 (0) | 8 (8)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 14 (16)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (11)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (5)
Proteinuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Menorrhagia (Reproductive system and breast disorders) | 0/1 (0) | 1/19 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (20)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 12 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (7) | 46 (96)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 26 (36)
Hirsutism (Skin and subcutaneous tissue disorders) | 0/1 (0) | 2/19 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 15 (36)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (15)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (33)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02451930/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT02451930/SAP_001.pdf